CLINICAL TRIAL: NCT04563351
Title: Randomized Clinical Trial on the Effectiveness of the Intraligamentary Anesthesia and Inferior Alveolar Nerve Block on Pain During Dental Treatment
Brief Title: Effectiveness of the Intraligamentary Anesthesia and Inferior Alveolar Nerve Block on Pain During Dental Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BB 174/18
Record Dates: First submitted 2020-09-11; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Dental Caries
Keywords: local anesthetic; dentistry; pain; techniques
MeSH Terms: conditions — Dental Caries; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional inferior alveolar nerve block (IANB) (Active Comparator): 37 patients received Inferior Alveolar Nerve Block (IANB) for dental treatment of mandibular posterior teeth.
  Interventions: Other: local anaesthetic techniques
- Intraligamentary Anesthesia (ILA) (Experimental): 35 patients received Intraligamentary Anesthesia (ILA) for dental treatment of mandibular posterior teeth.
  Interventions: Other: local anaesthetic techniques

INTERVENTIONS:
Other: local anaesthetic techniques — The patients were anesthetized with two different local anaesthetic techniques.

SUMMARY:
Objective: To compare the effectiveness and complications of intraligamentary anesthesia (ILA) with conventional inferior alveolar nerve block (IANB) during injection and dental treatment of mandibular posterior teeth.

Materials and Methods: In this randomized, prospective clinical trial, 72 patients (39 males, 33 females) patients scheduled for dental treatment of mandibular posterior teeth, were randomly allocated to ILA group (n=35) received ILA injection or IANB group (n=37) received the conventional IANB. Our primary outcome was to assess pain during the injection as well as pain and stress (discomfort) during dental treatment, using the Numeric Rating Scale (NRS) from 0 to 10 (0 = no pain, 10= the worst pain imaginable). Whereas; recording 24 hours postoperative complications were our Secondary outcomes.

DETAILED DESCRIPTION:
MATERIALS AND METHODS This prospective randomized comparative clinical trial was conducted in the integrated clinical course in the dental school of the University of Greifswald, Germany after the approval of the local ethics committee of the medical faculty in Greifswald (No. BB 174/18) in a period from December 2018 to June 2019. The sample size calculation using "G*power version 3.1" (Heinrich-Heine-University / Germany) was based on the following estimates: T-test for means (difference between two independent means), effect size 0.7, α error 0.05 and power (1-ß error) 0.9. It resulted in a samples size of 36 patients in each of the two groups (IANB & ILA).

Inclusion and Exclusion Criteria The patients requiring regular dental in permanent mandibular posterior teeth under local anesthesia were recruited with an age range of 18 to 50 years. Patients were not included if they had a clinical or radiographic sign of acute abscess, pus or peri-radicular pathology. Also patients with a systemic disease requiring special considerations during their dental treatment or patients with contra-indications for any of the components of the anesthetic solution (allergy to articaine, epinephrine, and sulfite) were excluded.

Clinical Treatment and Outcome Computer-generated randomization technique was applied to allocate the participants to one of the both study groups (ILA vs. IANB). The intensity of pain as well as stress during the injection of the local anesthesia and during the dental procedure was assessed by using the Numeric Rating Scale (NRS 0-10). The anesthesia was performed by the clinical instructors of the course being dental practitioners (GDPs) or by dental students in the 4th and 5th academic year in the integrated clinical course in the dental school of the University of Greifswald and recorded as dentist or student. The distributions of different experience level of clinical instructors, dental students in 4th and 5th year were considered. For the inferior alveolar nerve block, the patient was placed comfortably in a supine position on the dental chair. The start of the anesthetic procedure was done without using topical anesthesia. The IANB injection was administered with cannulas of 38 mm in length and a gauge of 0.4 mm (Sopira Carpule, Heraeus Kulzer GmbH Hanau, Germany). The patients were anesthetized with Ultracain DS Forte 1:100.00 (Sanofi Aventis, Germany), the active ingredient being articaine in 1.7 ml ampules (1 ml equal to 40 mg articaine hydrochloride and 0.012 mg epinephrine hydrochloride, which is included as a vasoconstrictor). Once the bone was contacted, 1.5 ml of anesthetic solution was injected slowly. Subsequently the needle was detached for approximately 1 cm and an addition of 0.3-0.5 ml of local anesthetic solution was injected to anesthetize the lingual nerve.

For the intraligamentary anesthesia, three different syringe systems were used with randomized selection: Softjet syringe (Henke-Sass Wolf, Tuttlingen, Germany), Citojet syringe (Sopira, Heraeus Kulzer GmbH Hanau, Germany), Ultrajet syringe (Sanofi-Aventis, Frankfurt am Main, Germany). The patients were also placed in a supine position and the dentist administered the ILA injection without using topical anesthesia with cannulas of 12 mm in length and a gauge of 0.30 mm (Sopira Carpule, Heraeus Kulzer GmbH Hanau, Germany). Also, Ultracain DS Forte 1:100.000 (Sanofi Aventis, Germany) was used from 1.7 ml ampules. The needle was navigated through the gingival sulcus with the bevel towards the alveolar bone and away from the root surface, at an angle of 30°-40° to the long axis of the tooth and 2- 3 mm into the periodontal ligament space between root and alveolar bone. For each root, 0.2 ml of local anesthetic was injected over at least 20 seconds according to Endo et al. (2008) as well as Bender and Taubenheim (2014).

ELIGIBILITY:
Inclusion Criteria:

* patients requiring regular dental in permanent mandibular posterior teeth under local anesthesia

Exclusion Criteria:

* Patients with a clinical or radiographic sign of acute abscess, pus or peri-radicular pathology
* Patients with a systemic disease requiring special considerations during their dental treatment
* Patients with contra-indications for any of the components of the anesthetic solution (allergy to articaine, epinephrine, and sulfite)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
The intensity of pain during the injection | immediately after the injection of LA
  The intensity of pain during the injection of the LA to be assessed by the patient using Numeric Rating Scale. The Numeric Rating Scale, (NRS 0-10; 0 representing no pain at all and 10 representing the worst pain imaginable) is a valid instrument to measure pain.
The intensity of pain during the dental treatment | immediately after the dental treatment
  The intensity of pain during the dental treatment to be assessed by the patient using Numeric Rating Scale. The Numeric Rating Scale, (NRS 0-10; 0 representing no pain at all and 10 representing the worst pain imaginable) is a valid instrument to measure pain.
The intensity of stress (discomfort) | immediately after the dental treatment
  The intensity of stress during the dental treatment to be assessed by the patient using Numeric Rating Scale. The Numeric Rating Scale, (NRS 0-10; 0 representing no discomfortable at all and 10 representing the maximal discomfortable very imaginable) is a valid instrument to measure stress (discomfort)

SECONDARY OUTCOMES:
Postoperative complications | 24 hours
  Recording any postoperative complications which could be occurred (Nerve injury or any other temporary irritations like the pain at the site of injection, signs of intravascular injection, lip-bit injury)

CONTACTS AND LOCATIONS:
Overall Officials: Christian splieth, PHD, Study Director — University Medicine of Greifswald
Locations (1):
- University Medicine of Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pradhan R, Kulkarni D, Shetty L. Evaluation of Efficacy of Intraligamentary Injection Technique for Extraction of Mandibular Teeth-A Prospective Study. J Clin Diagn Res. 2017 Jan;11(1):ZC110-ZC113. doi: 10.7860/JCDR/2017/22204.9302. Epub 2017 Jan 1. PMID 28274058
- [Result] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Result] Siegel K, Schrimshaw EW, Kunzel C, Wolfson NH, Moon-Howard J, Moats HL, Mitchell DA. Types of dental fear as barriers to dental care among African American adults with oral health symptoms in Harlem. J Health Care Poor Underserved. 2012 Aug;23(3):1294-309. doi: 10.1353/hpu.2012.0088. PMID 24212175
- [Result] Bahl R. Local anesthesia in dentistry. Anesth Prog. 2004;51(4):138-42. No abstract available. PMID 15675263
- [Result] Shabazfar N, Daublander M, Al-Nawas B, Kammerer PW. Periodontal intraligament injection as alternative to inferior alveolar nerve block--meta-analysis of the literature from 1979 to 2012. Clin Oral Investig. 2014;18(2):351-8. doi: 10.1007/s00784-013-1113-1. Epub 2013 Sep 29. PMID 24077785
- [Result] Kaufman E, Weinstein P, Milgrom P. Difficulties in achieving local anesthesia. J Am Dent Assoc. 1984 Feb;108(2):205-8. doi: 10.14219/jada.archive.1984.0470. No abstract available. PMID 6584494
- [Result] Pogrel MA. Permanent nerve damage from inferior alveolar nerve blocks--an update to include articaine. J Calif Dent Assoc. 2007 Apr;35(4):271-3. PMID 17612365
- [Result] Marniemi J, Parkki MG. Radiochemical assay of glutathione S-epoxide transferase and its enhancement by phenobarbital in rat liver in vivo. Biochem Pharmacol. 1975 Sep 1;24(17):1569-72. doi: 10.1016/0006-2952(75)90080-5. No abstract available.
- [Result] Kämmerer PW, Palarie V, Schiegnitz E, Ziebart T, Al-Nawas B, Daubländer M. Clinical and histological comparison of pulp anesthesia and local diffusion after periodontal ligament injection and intrapapillary infiltration anaesthesia. J Pain Relief. 2012;1(10.4172):2167-0846.
- [Result] Walton RE, Garnick JJ. The periodontal ligament injection: histologic effects on the periodontium in monkeys. J Endod. 1982 Jan;8(1):22-6. doi: 10.1016/S0099-2399(82)80312-9. No abstract available. PMID 6948904
- [Result] Dreyer WP, van Heerden JD, de V Joubert JJ. The route of periodontal ligament injection of local anesthetic solution. J Endod. 1983 Nov;9(11):471-4. doi: 10.1016/S0099-2399(83)80161-7. No abstract available. PMID 6586974
- [Result] Kammerer PW, Adubae A, Buttchereit I, Thiem DGE, Daublander M, Frerich B. Prospective clinical study comparing intraligamentary anesthesia and inferior alveolar nerve block for extraction of posterior mandibular teeth. Clin Oral Investig. 2018 Apr;22(3):1469-1475. doi: 10.1007/s00784-017-2248-2. Epub 2017 Oct 15. PMID 29034443
- [Result] Meechan JG. Intraligamentary anaesthesia. J Dent. 1992 Dec;20(6):325-32. doi: 10.1016/0300-5712(92)90018-8. PMID 1452871
- [Result] Endo T, Gabka J, Taubenheim L. Intraligamentary anesthesia: benefits and limitations. Quintessence Int. 2008 Jan 1;39(1):e15-25. PMID 18551207
- [Result] Kammerer PW, Schiegnitz E, von Haussen T, Shabazfar N, Kammerer P, Willershausen B, Al-Nawas B, Daublander M. Clinical efficacy of a computerised device (STA) and a pressure syringe (VarioJect INTRA) for intraligamentary anaesthesia. Eur J Dent Educ. 2015 Feb;19(1):16-22. doi: 10.1111/eje.12096. Epub 2014 Mar 20. PMID 24646115
- [Result] Reed KL, Malamed SF, Fonner AM. Local anesthesia part 2: technical considerations. Anesth Prog. 2012 Fall;59(3):127-36; quiz 137. doi: 10.2344/0003-3006-59.3.127. PMID 23050753
- [Result] Dumbrigue HB, Lim MV, Rudman RA, Serraon A. A comparative study of anesthetic techniques for mandibular dental extraction. Am J Dent. 1997 Dec;10(6):275-8. PMID 9590915
- [Result] Prama R, Padhye L, Pawar H, Rajput N. Efficacy of Intraligamentary Injections as a Primary Anesthetic Technique for mandibular molars & a comparison with inferior alveolar nerve block. Indian Journal of Multidisciplinary Dentistry. 2013 Aug 1;3(4).
- [Result] Malamed SF. Handbook of local anesthesia. Elsevier Health Sciences; 2004 Jun 8.
- [Derived] Youssef BR, Sohnel A, Welk A, Abudrya MH, Baider M, Alkilzy M, Splieth C. RCT on the effectiveness of the intraligamentary anesthesia and inferior alveolar nerve block on pain during dental treatment. Clin Oral Investig. 2021 Aug;25(8):4825-4832. doi: 10.1007/s00784-021-03787-x. Epub 2021 Feb 1. PMID 33527192